CLINICAL TRIAL: NCT00897806
Title: Feasibility of Measuring Gene Expression Patterns Using Tissue Acquisition of Primary Stage 3 & 4 Epithelial Ovarian Cx or Primary Peritoneal Cx & Gene Expression Array Technology for Predicting Paclitaxel Chemotherapy
Brief Title: Identifying Genetic Markers That Predict Response to Paclitaxel in Patients With Newly Diagnosed Stage III or Stage IV Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Terminated | Type: Observational
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID00-408; P50CA083639 (NIH); P30CA016672 (NIH); MDA-ID-00408 (Other: UT MD Anderson Cancer Center); CDR0000355794 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Microarray Analysis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples undergo transcriptional profiling using cDNA microarrays.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Genetic Markers
  Interventions: Genetic: Microarray analysis; Other: Laboratory biomarker analysis

INTERVENTIONS:
Genetic: Microarray analysis
Other: Laboratory biomarker analysis

SUMMARY:
RATIONALE: DNA analysis of tumor tissue from patients with cancer may help doctors predict how patients respond to treatment and plan the best treatment.

PURPOSE: This laboratory study is identifying genetic markers that predict response to paclitaxel in patients with newly diagnosed stage III or stage IV ovarian epithelial cancer or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Identify genetic markers of paclitaxel chemosensitivity and/or chemoresistance, using gene expression arrays, in patients with newly diagnosed stage III or IV ovarian epithelial cancer or primary peritoneal cancer treated with single-agent weekly paclitaxel followed by paclitaxel in combination with carboplatin.
* Correlate RNA expression levels with clinical response in patients treated with this regimen.

Secondary

* Determine the response rate in patients treated with this regimen.
* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Compare transcriptional profiles of primary tumors vs tissue obtained at second-look surgery in patients treated with this regimen.
* Identify differential expression between pre- and post-treatment tissue in patients treated with this regimen.

OUTLINE: This is a pilot study.

Pre- and post-chemotherapy tumor samples undergo transcriptional profiling using cDNA microarrays to identify gene overexpression. The gene expression profiles of paclitaxel-sensitive tumors are compared with those that are paclitaxel resistant to identify gene markers that are associated with response to paclitaxel.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly diagnosed histologically confirmed advanced stage (III & IV) epithelial ovarian cancer, fallopian tube or peritoneal cancer. --OR-- Patients with a suspected malignancy who are unsuitable candidates for surgery (i.e., those with medical co-morbidities, massive effusions, or tumor burden such that an optimal resection is unlikely) who undergo a core biopsy that is positive for malignancy.
2. Patients who have undergone tumor reduction must have either stage III suboptimal (> 2 cm residual) disease or stage IV disease.
3. Patients may have had no prior chemotherapeutic regimen.
4. Zubrod performance status of 0, 1, or 2.
5. Patients must have recovered from effects of recent surgery. They should be free of significant infection.
6. Patients must have adequate: Bone marrow function: WBC >/= than 3,000/microlitre, platelets > 100,000/microlitre, absolute neutrophil (ANC) count >/= than 1.5/microlitre. Renal function: Creatinine </= 1.5 mg%. Hepatic function: Bilirubin </= 1.5 mg/dl, SGOT and alkaline phosphatase </= 3 X institutional normal.
7. Patients must have adequate: Neurologic function: Pre-existing peripheral neurologic toxicity is allowed but limited to parasthesia and decreased vibratory sense without motor weakness. Intermittent constipation managed with laxatives is allowed, without evidence of bowel obstruction. Psychiatric function: Functions independently without evidence of delirium, confusion, suicidal ideation, or untreated depression.
8. Patients who have signed an approved informed consent.

Exclusion Criteria:

1. Patients with borderline or grade 1 (low grade) tumors.
2. Patients who have received any prior cytotoxic chemotherapy or radiotherapy.
3. Patients with septicemia, severe infection, acute hepatitis, or gastrointestinal bleeding at the time of protocol entry.
4. Patients with unstable angina or those who have had a myocardial infarction within the past six months. Patients with evidence of abnormal cardiac conduction (e.g., bundle branch block, heart block, etc.) are eligible if their disease has been stable for the past six months.
5. Patients whose circumstances do not permit completion of the study or the required follow-up.
6. Patients with a history of another malignancy within 5 years. Patients who have had a prior malignancy but remain continuously free of recurrent or persistent disease for more than 5 years may be entered in the study after consultation with the study chair.
7. Patients with significant pre-existing cardiac disease (NYHA class III-IV) will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed Stage III or Stage IV Ovarian Epithelial Cancer or Primary Peritoneal Cancer.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2002-02; Primary Completion 2006-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Genetic markers of paclitaxel chemosensitivity and/or chemoresistance | 2 years
Correlation of RNA expression levels with clinical response | 2 years

SECONDARY OUTCOMES:
Response rate to weekly paclitaxel in chemotherapy naive patients | Every 3 months post treatment
  Resonse measured by clinical assessments every 3 months post treatment.
Progression-free survival | Every 3 months post treatment
  Influence of weekly paclitaxel followed by paclitaxel in combination with carboplatin on progression-free survival by clinical assessments every 3 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: David M. Gershenson, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org